CLINICAL TRIAL: NCT07401745
Title: Combination Treatment of Occlusal Splint Appliance and Granisetron Injection Into the Masseter Muscle for Managing of Myofascial Pain Related to Temporomandibular Disorders: A Randomized Controlled Parallel-arm Clinical Trial
Brief Title: Occlusal Splint Combined With Granisetron Injection for Managing Myofascial Pain Related to Temporomandibular Disorders
Acronym: TMD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sarah Elmaghraby, Lecturer, Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University, Mansoura, Egypt., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.25.10.27
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: TMD; TMD/Orofacial Pain; Temporomandibular Disorder (TMD)
Keywords: TMD; temporomandibular disorder; orofacial pain; myofascial pain; granisetron; lidocaine; occlusal splint
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain | interventions — Granisetron; Lidocaine; Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Granisetron (Granitryl 1 mg/ml, ampules, EGYPHARMA-Egypt) will be used in group II, while lidocaine (2%lidocaine hydrochloride, pharco, egypt) will be used in group III. The most painful tender-points to palpation of the masseter muscle will be marked, maximum 3 per muscle. The injected volume into each tender-point was 0.5 mL. Thus the maximum dose of granisetron a patient could receive was 3 mg per treatment. As for lidocaine the same amount as granisetron was injected the same way, maximum safe amount injected will be below the maximum safe dosage (mg/kg) of lidocaine. The injections were made perpendicular to the skin surface over the chosen tender-point with an angle of 90° using a 19-mm long needle (diameter 0.4 mm) from a 2-mL syringe. The solution was administered into each tender-point as a single shot during 10 s. In order to en sure intramuscular administration. The injections were repeated after 1week in the most painful tender-points at that time.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Only occlusal splint group (Active Comparator): This group will receive occlusal splint therapy only.
  Interventions: Device: occlusal splint
- Occlusal splint and granisetron injection group (Experimental): This group will receive occlusal splint therapy in addition to a single dose of granisetron that will be administered via intramuscular injection at a dose of 0.5 mL.
  Interventions: Drug: Granisetron; Device: occlusal splint
- Occlusal splint and lidocaine injection group (Experimental): This group will receive occlusal splint therapy in addition to a single dose of lidocaine that will be administered via intramuscular injection at a dose of 0.5 mL.
  Interventions: Drug: lidocaine; Device: occlusal splint

INTERVENTIONS:
Drug: Granisetron — Granisetron (Granitryl 1 mg/ml, ampules, EGYPHARMA-Egypt)
  Arms: Occlusal splint and granisetron injection group
Drug: lidocaine — lidocaine (2%lidocaine hydrochloride, pharco, egypt)
  Arms: Occlusal splint and lidocaine injection group
Device: occlusal splint — Specially designed mouth guards that change the occlusal relationship of maxillary and mandibular teeth to improve the alignment of the tooth contact, with the aim of relieving temporomandibular pain.

SUMMARY:
The goal of this clinical trial is to evaluate whether a combination of occlusal splint therapy and granisetron injection into the masseter muscle is effective in managing myofascial pain related to temporomandibular disorders (TMD). The study will also compare this combination treatment to occlusal splint therapy alone and to occlusal splint therapy combined with lidocaine injection.

The main questions this study aims to answer are:

* Does adding granisetron injection to occlusal splint therapy reduce myofascial pain more effectively than occlusal splint therapy alone?
* How does granisetron injection compare to lidocaine injection when combined with occlusal splint therapy?
* Does the combination treatment improve mandibular movement and reduce joint clicking?
* Are there any local or systemic side effects associated with granisetron or lidocaine injections?

Researchers will compare three groups to evaluate treatment effectiveness:

* Occlusal splint therapy alone
* Occlusal splint therapy plus granisetron injection
* Occlusal splint therapy plus lidocaine injection

Participants will:

* Wear an occlusal splint as part of their treatment
* Attend follow-up visits after 1 week, 1 month, 3 months, and 6 months

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 -45 years.
* Diagnosis of myofascial pain according to the Research Diagnostic Criteria for TMD Axis I (RDC/TMD).
* Pain upon digital palpation of the masseter and/or the temporalis muscles.
* Patients with disc displacement with or without reduction in any of the TMJs.
* Co-operative patients.

Exclusion Criteria:

* Diagnosed systemic muscular or joint diseases (e.g. fibromyalgia, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis).
* Whiplash associated disorder.
* Neuropathic pain or neurological disorders (e.g. myasthenia gravis, orofacial dystonia).
* History of psychiatric disorders.
* Pain of dental origin.
* Use of muscle relaxants or any medication that might influence the response to pain.
* Pregnancy or lactation.
* Known hypersensitivity to granisetron or lidocaine

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Preoperatively and 1 week, 1month, 3 months and 6 months post operatively.
  Pain intensity will be assessed using a Visual Analogue Scale (VAS), where 0 represents no pain and 10 represents the worst imaginable pain. Participants will mark their pain at rest and during jaw movements
Presence or absence of a clicking sound | Preoperatively and 1 week, 1month, 3 months and 6 months post operatively.

SECONDARY OUTCOMES:
Electrical activity of muscles | Preoperatively and 6 months postoperatively.
  Electromyography will be acomplished using MyoWise (Myowise EMG/device, cometa srl manufacturing, Italy) device which is a surface electromyography (sEMG) system designed to record and analyze the electrical activity of muscles- Page 3 of 5 [DRAFT] during rest and function. It utilizes adhesive surface electrodes to detect muscle action potentials, which are amplified, filtered, and displayed as real-time signals on a connected computer or tablet. The system provides quantitative data on muscle activation patterns, amplitude, and timing, allowing assessment of neuromuscular activity and coordination.
Maximum interocclusal opening | Preoperatively and 1 week, 1month, 3 months and 6 months post operatively.
Range of lateral mandibular movement | Preoperatively and 1 week, 1month, 3 months and 6 months post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Elmaghraby, Lecturer, Principal Investigator — Faculty of Dentistry, Mansoura University, Mansoura, Egypt.
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No